CLINICAL TRIAL: NCT03146000
Title: Effect of Topical Lidocaine-prilocaine Cream Versus Rectal Meloxicam Suppository on Relief of Post-episiotomy Pain: A Randomized Clinical Trial
Brief Title: Lidocaine-prilocaine Cream Versus Rectal Meloxicam on Relief of Post-episiotomy Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEP
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine-prilocaine (Experimental): women will receive 5 mg lidocaine-prilocaine cream topically on the episiotomy line
  Interventions: Drug: lidocaine-prilocaine cream
- meloxicam (Active Comparator): women will receive one 15 mg meloxicam rectal suppository
  Interventions: Drug: meloxicam rectal suppository

INTERVENTIONS:
Drug: lidocaine-prilocaine cream — topical cream
  Arms: lidocaine-prilocaine
Drug: meloxicam rectal suppository — suppository
  Arms: meloxicam

SUMMARY:
Postpartum perineal pain is a very common complaint. It can have negative consequences for mother and child including disability in daily functioning for the mother; for example, it can interfere in taking care of her infant and in breastfeeding. Early pain management is thus relevant to provide relief and prevent chronicity.

Perineal pain is particularly common following childbirth. Macarthur 2004, in a prospective cohort study involving 447 women in Canada, reported an incidence of perineal pain, in the first day after birth, of 75% in women with an intact perineum

ELIGIBILITY:
Inclusion Criteria:

1. Primiparas
2. Normal vaginal delivery
3. Mediolateral episiotomy
4. Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

1. Patients who had postpartum hemorrhage
2. Patients who had manual removal of the placenta
3. Patients with contraindications to non steroidal drugs
4. Patients with a multiple perineal lacerations

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
The mean difference of visual analog scale after delivery | immediately
  the scale is graded from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No